CLINICAL TRIAL: NCT00351793
Title: A Clinical Trial Follow-up Study of the Genesis II Posterior Stabilized Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Ross Leighton (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Ross Leighton, Orthopedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: CDHA-RL-004
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Knee Prosthesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Combined Deformity <30 degrees
  Interventions: Device: Knee Implant
- Combined Deformity >30 degrees
  Interventions: Device: Knee Implant

INTERVENTIONS:
Device: Knee Implant — Total knee replacement with Genesis II posterior stabilized knee

SUMMARY:
The purpose of this study is to look at the outcomes of the GENESIS II Posterior Stabilized Total Knee Replacement.

ELIGIBILITY:
Inclusion Criteria:

* A combined deformity of <30 degrees = group 1
* A combined deformity of >30 degrees = group 2
* Patient is willing to consent to participate in the study
* Patient is available for follow-up through at least 2 years but preferably 5 years
* Patient has met acceptable preoperative medical clearance and is free of or treated for medical conditions that would pose excessive operative risk
* Patients who are fluent in English and are able to understand their role in a clinical trial

Exclusion Criteria:

* Active, local infection or systemic infection
* Fibromyalgia patients
* Patients whom, as judged by the surgeon, are not capable of understanding the informed consent or the requirements of the protocol and or are reasonably unlikely to be compliant with the prescribed routine and the follow-up evaluation schedule

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Total knee replacement candidates
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2003-01; Primary Completion 2018-12 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness and Safety | 5 years
  Will evaluate effectiveness and safety during a 5 year period via analysis of the Knee Society Score, revision status, and radiographic evaluation

SECONDARY OUTCOMES:
Knee Society Clinical Rating | Pre-op, 6 months, 1 year, 2 years, 5 years
Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC) | Pre-op, 6 months, 1 year, 2 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ross K Leighton, MD, FRCS(C), Principal Investigator — Capital Health, Canada
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada